CLINICAL TRIAL: NCT04186234
Title: Prospective Study of Stereotactic Body Radiation Therapy as Bridging Therapy for Hepatocellular Carcinoma Patients on Waiting List for Liver Transplantation
Brief Title: SBRT for Liver Cancer Before Liver Transplantation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Victor H.F. Lee, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 15-191
Record Dates: First submitted 2019-12-01; First posted 2019-12-04 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Liver Cancer; Liver Transplant Disorder
Keywords: Liver cancer; Stereotactic body radiation therapy; Bridging therapy; Liver transplantation
MeSH Terms: conditions — Liver Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Stereotactic body radiation therapy as bridging therapy before liver transplantation for hepatocellular carcinoma
Masking Description: Inapplicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stereotactic body radiation therapy (Experimental): Stereotactic body radiation therapy of 35 to 50 Grays in 5 fractions over 5 to 14 days.
  Interventions: Radiation: Stereotactic body radiation therapy

INTERVENTIONS:
Radiation: Stereotactic body radiation therapy — Stereotactic body radiation therapy of 30 to 50 Grays in 5 fractions before liver transplantation

SUMMARY:
Hepatocellular carcinoma (HCC) is the second commonest cause of cancer death worldwide. It is the third leading cause of cancer death in Hong Kong. Liver transplantation (LT) is the curative treatment of choice for HCC as it has the advantage of removing the tumour and also the premalignant cirrhotic liver. Milan (solitary tumour <5cm, or up to 3 tumours, each <3cm) and University of California San Francisco (UCSF) criteria (solitary tumour ≤6.5cm, up to 3 tumours with none >4.5cm, and total tumour diameter ≤8cm) provide the benchmark requirements for LT, at which a 5-year survival of >70% and recurrence rate ranging from 5-15% can be achieved. However, organ shortage and waiting time for liver grafts remain the greatest obstacles for deceased donor liver transplantation (DDLT). It has been reported that the waiting list dropout rate is 7 to 11% at 6 months and 38% at 12 months. Several therapeutic procedures including transarterial chemoembolisation (TACE) and stereotactic body radiation therapy (SBRT) have been studied as bridging therapy before DDLT, aiming at reducing waiting list dropout rate and recurrence after LT, and improving post-transplant survival.

The investigators have carried out a prospective study on HCC patients treated with bridging SBRT before LT. The investigators used dual tracer (18F-fluorodeoxyglucose [FDG] and 11carbon-acetate [ACC]) positron-emission tomography with integrated computed tomography (PET-CT) and magnetic resonance imaging with gadoxetate disodium as baseline and subsequent imaging assessment before and after SBRT, hoping the PET-CT can help better identify those who benefit from SBRT and to prioritise those with poor response so that they can be better channeled to LT.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the second commonest cause of cancer death worldwide. It is the third leading cause of cancer death in Hong Kong. Liver transplantation (LT) is the curative treatment of choice for HCC as it has the advantage of removing the tumour and also the premalignant cirrhotic liver. Milan (solitary tumour <5cm, or up to 3 tumours, each <3cm) and University of California San Francisco (UCSF) criteria (solitary tumour ≤6.5cm, up to 3 tumours with none >4.5cm, and total tumour diameter ≤8cm) provide the benchmark requirements for LT, at which a 5-year survival of >70% and recurrence rate ranging from 5-15% can be achieved. However, organ shortage and waiting time for liver grafts remain the greatest obstacles for deceased donor liver transplantation (DDLT). It has been reported that the waiting list dropout rate is 7 to 11% at 6 months and 38% at 12 months. Several therapeutic procedures including transarterial chemoembolisation (TACE) and stereotactic body radiation therapy (SBRT) have been studied as bridging therapy before DDLT, aiming at reducing waiting list dropout rate and recurrence after LT, and improving post-transplant survival. TACE is the most widely used bridging therapy with tumour necrosis rate of 25-57% on explant pathology.

However it is largely only feasible in patients with Child-Pugh Class A status. SBRT, through the delivery of extremely conformal tumouricidal radiation in a few fractions (usually ≤5) under real-time liver and tumour motion monitoring, is more fashionable. Prospective studies have shown a higher local control rate of 87-100% at 1 year, an overall survival of 60-69% at 2 years after SBRT for unresectable HCC with minimal radiation-induced liver disease (RILD) compared to TACE. Studies have also been made on the use of SBRT as bridging therapy. Computed tomography (CT) and magnetic resonance imaging (MRI) have traditionally been used to diagnose and monitor treatment response for HCC. Their sensitivity and specificity are comparable for lesions >2cm. MR imaging provides higher soft tissue contrast and addition of liver-specific contrast agent (gadoxetate disodium, Primovist) further improves detection of 1-2cm tumours, demonstrating 92.1% accuracy based on the Milan and UCSF guidelines. However MRI is subject to significant motion artefacts during scanning. 18F-fluorodeoxyglucose (FDG) PET-CT has been extensively studied in HCC staging and treatment response monitoring. Unfortunately, FDG PET-CT is only capable of detecting the more poorly-differentiated component of HCC. It was first found in Hong Kong in 2003 that 11carbon-acetate (ACC) can detect the more well-differentiated component and both FDG and ACC as dual tracers have an incremental value of diagnosing extra-hepatic metastases in comparison to FDG alone. It was further proven by our hepatobiliary surgical team that ACC improved overall sensitivity of diagnosis in the pre-transplant cohort.

Few studies have looked at PET-CT for treatment response evaluation. A previous study has shown that cohorts with higher standardised uptake value (SUV) ratios have higher responses to external radiotherapy than lower SUV ratios cohort. However, the population was small and the treatment regimens were inhomogeneous. Use of FDG PET-CT has been promising in assessing treatment response after TACE and Y-90 microspheres selective internal radiation therapy (SIRT). However, there are very few publications on dual tracer PET-CT scan to evaluate tumour response after SBRT.

In view of the above, the investigators have carried out a prospective study on HCC patients treated with bridging SBRT before LT. The investigators used dual tracer (FDG and ACC) positron-emission tomography with integrated computed tomography (PET-CT) and MRI with gadoxetate disodium as baseline and subsequent imaging assessment before and after SBRT, hoping the dual tracer PET-CT and MRI with gadoxetate disodium can help better identify those who benefit from SBRT and to prioritise those with poor response so that they can be better channeled to LT.

ELIGIBILITY:
Inclusion criteria:

1. Patients must have histologically or radiologically confirmed HCC. For radiological diagnosis of HCC, a contrast-enhanced computed tomography or magnetic resonance imaging is mandatory to demonstrate the early arterial enhancement in arterial phase and contrast washout in the porto-venous phase on the imaging
2. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorisation (e.g. Health Insurance Portability and Accountability Act in the US, Euripean Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations
3. HCC lesions with Milan criteria or University of San Francisco criteria for LT
4. Be >/= 18 years of age on day of signing informed consent
5. Have a performance status of 0 or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
6. A stage C or earlier HCC based on Barcelona Clinic Liver Cancer (BCLC) staging system.
7. A Child-Pugh of 8 or less.
8. Demonstrate adequate organ function as defined in Inclusion Criteria 9, all screening labs should be performed 28 days prior to study registration up to first dose of study drug.
9. Adequate serum hematological functions defined as:

   * Absolute neutrophil count (ANC) ≥1.0 x 10^9/l
   * Platelet ≥20 x 10^9/l
   * Haemoglobin ≥8 g/dL

   Adequate serum biochemistry functions defined as:
   * Serum bilirubin ≤5.0 x institutional upper limit of normal (ULN). <<This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinaemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.>>
   * AST (SGOT)/ALT (SGPT) ≤6 x institutional upper limit of normal
   * Albumin ≥25g/litre
   * Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Males:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

   Females:

   Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
10. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 2.0 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants. Activated Partitional Thromboplastin Time (aPTT) ≤ 2.0 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
11. Female subject of childbearing potential should have a negative urine or serum pregnancy within 24 hours of study enrollment up to administration of the dose of study drug. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 31 weeks after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilised or have not been free from menses for > 1 year. The following age-specific requirements apply:

    * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinising hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilisation (bilateral oophorectomy or hysterectomy).
    * Women ≥50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilisation (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
13. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 31 weeks after the last dose of study therapy.
14. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
15. Must have a life expectancy of at least 12 weeks.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment or 5 half-lives, whichever is shorter.
2. Has a diagnosis of severe active scleroderma, lupus, other rheumatologic or autoimmune disease within the past 3 months before study recruitment. Patients with a documented history of clinically severe autoimmune disease or a syndrome requiring systemic steroids or immunosuppressive agents will not be allowed on this study. Subjects with vitiligo or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections are not excluded from the study. Subjects with hypothyroidism stable on hormone replacement are not excluded from this study.
3. Has had a prior monoclonal antibody, immunotherapy or immune checkpoint inhibitors before recruitment into this study.
4. Has had prior chemotherapy or targeted small molecule therapy (including sorafenib, lenvatinib, or other anti-vascular endothelial growth factor inhibitor) before recruitment into this study.
5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, indolent lymphomas, or in situ cervical cancer that has undergone potentially curative therapy
6. Has a history of prior solid organ transplants with or without any episodes of graft-versus-host disease.
7. Has a history of allogeneic bone marrow transplantation and peripheral stem cell rescue, with or without any episodes of graft-versus-host disease.
8. Has known extra-hepatic metastases.
9. Has known carcinomatous meningitis (also known as leptomeningeal carcinomatosis)
10. Has an active infection requiring intravenous systemic therapy or hospital admission.
11. Has a history or current evidence of any condition, therapy, or laboratory abnormality, including psychiatric or substance abuse disorder, that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 31 weeks after the last dose of trial treatment.
13. Untreated hepatitis B infection. Patients with chronic hepatitis B infection (defined as HBsAg positive) are eligible if they have started anti-viral therapy for at least 1 month and is continuing anti-viral treatment throughout the whole duration of this study.
14. Has experienced Grade 4 toxicity on treatment with prior radiation if done before.
15. Prior systemic therapy utilising an anti CTLA-4 or PD-1/PD-L1 agent or other forms of immunotherapy.
16. Has had prior radiation therapy (defined as >0.5Gy) to the area planning to be treated with SBRT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 36 months
  Progression-free survival
Best objective response | 36 months
  Best objective response

SECONDARY OUTCOMES:
Overall survival | 36 months
  Overall survival

OTHER OUTCOMES:
Toxicity profile | 36 months
  Toxicity profile
Changes in Child-Pugh status | 36 months
  Changes in Child-Pugh status (A, B, or C) after stereotactic body radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Victor Lee, MD, Principal Investigator — Department of Clinical Oncology, The University of Hong Kong, Hong Kong
Locations (1):
- Department of Clinical Oncology, Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be routinely available to other researchers unless if our site is invited by other parties for individual patient data meta-analysis